CLINICAL TRIAL: NCT04430374
Title: Qatar Cardiovascular COVID-19 Registry
Brief Title: Registry for a Cardiovascular Patient Who COVID-19 Infection in Qatar and Gulf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. JASSIM MOHD. AL SUWAIDI, Senior Cardiologist, Hamad Medical Corporation
Other Study IDs: MRC-05-113
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interverntion — No intervention will be done, registry only

SUMMARY:
The novel coronavirus, severe acute respiratory syndrome coronavirus 2, that causes coronavirus disease 2019 (COVID -19), is highly contagious in the community and has resulted in a global pandemic. This infection has a special implication on the patient who complains from cardiac disease or acute cardiovascular condition and may result in cardiovascular complications such as myocardial infarction. For this end, we target to study this group of patient, who has a cardiac disease with COVID-19 in Qatar, in addition, the acute myocardial infarction with COVID-19 from the Gulf countries and collect all the related data to come with a comprehensive view about those patients.

DETAILED DESCRIPTION:
The primary objective of this registry is to create a database of patients who present with acute cardiovascular and are found to be COVID -19 positive (by PCR). The registry will consist of four arms (1) Retrospective data for all patients since the COVID-19 appear in Qatar unit the date of submission the protocol (2) Prospective data starting from the date of submission of this protocol and forward until end of December 2020 (3) Retrospective data for all cardiac patients hospitalizations in the COVID period of this year 2020 will be compared to previous years to report the trends of acute cardiovascular conditions in the COVID era to previous data, as a lot of countries documented decrease in the incidence. (4) retrospective data for acute MI and found to be COVID-19 until this protocol amendment from participating hospitals in the Gulf region to be compared with Acute MI from Qatar who collected in arm 1. The registry will consist of patients admitted with AMI who were already having active COVID-19 infection or were incidentally found to have COVID-19 by PCR. Additionally, prospective data from the data of this protocol amendment until the end of December 2020. This arm target to (a) increases the number of the collected patient for Acute MI with COVID-19category due to the small number in Qatar alone. (b) give the opportunity for Qatar to lead a multicenter project to serve in a hot topic, in particular, the data collection and analysis will be in Qatar. (c) allow releasing a publication for one cardiovascular center (Qatar only) and multi-cardiovascular center (all the Gulf), a multi-center publication about this issue could be rare on the worldwide level, and finally, (d) to increase the accuracy of the data analysis due to larger data size and comparing more than one site together.

Secondary plan to compare our patients' populations and outcomes with that of other international registries such as the NACMI(US registry). The NACMI registry is a rapid collaboration of multinational societies and medical institutions with a pragmatic study design to encourage widespread participation that will enable the development of data-driven guidelines and therapies.

The subject will be patients with confirmed or suspected COVID -19 infection with the acute cardiovascular conditions at the time of presentation to the hospital or that developed while in the hospital. All the history, laboratory results, current admission data, medication, angiogram, or intervention procedure (if underwent), and any other relevant data will be collected. All the patients who are applicable for this registry and meet the inclusion criteria will be involved so the final number of the subject is not specified. All patients with the acute coronary syndrome, out of hospital cardiac arrest and arrhythmias who are found to be COVID positive and required hospitalization will be included.

The following data variables will be collected as covariates of interest: baseline demographic and clinical characteristics, laboratory data, and pattern of ST-segment elevation (diffuse, focal, with or without ST-segment depression and/or PR -segment depression) transthoracic echocardiography or point-of-care ultrasound findings, commonly used time to treatment metrics in STEMI care (door -to -balloon or door -to -needle times), angiographic characteristics, and adjunctive pharmacological and device therapies including mechanical circulatory support (MCS ).

Implications for COVID -19 positive patients Observational registries have gained traction in cardiovascular medicine as they provide important information, including benefits and potential complications of different treatments or procedures. [12] For example, consecutive enrollment of patients with well -defined entry criteria in the Chest pain -MI Registry has been a reliable source for outcome-based, a quality improvement on high -risk STEMI/NSTEMI patients. [13] Immediate access to actionable data is particularly relevant to the current expanding COVID -19 pandemic which is disproportionally affecting cardiovascular patients and healthcare workers. [14] At present, there is no data-driven consensus on the management of patients with confirmed or suspected COVID -19 infection who present with ST-segment elevation on ECG. [11,15,16] The NACMI registry will be beneficial in identifying etiology, patterns of myocardial injury, developing a risk model for cardiac complications, understanding short and long -term major adverse cardiac events, and designing clinical trials testing different treatment modalities. Therefore, the registry will include both COVID -19 positive patients and PUI with acute cardiovascular conditions. A comparison of PUI subsequently confirmed positive to those subsequently confirmed negative will provide a unique insight into the pathophysiologic mechanism of STEMI from COVID -19, including myocarditis and prothrombotic states. Comparison of patients enrolled in NACMI to propensity-matched non -COVID STEMI controls for 1 year prior will provide critical information regarding etiology, treatment strategies and clinical outcomes in the COVID -19 pandemic. As testing for COVID -19 becomes more rapid, this decision -making process is expected to evolve. Additionally, it has been reported that overall STEMI volumes have decreased in the COVID -19 era, without a clear understanding of the reasons. [17,18] It may be that patients are delaying their presentation to the hospital, potentially leading to the need for mechanical circulatory support in the acute setting, mechanical complications of STEMI, sudden death or an increased heart failure population. Additionally, if patients are presenting later in their clinical course, NACMI registry data will allow practitioners to improve care models to improve time to treatment in this unique era.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who admitted to the heart hospital or any other hospital with acute cardiovascular condition.
2. Patient with confirming or suspicious of COVID-19 infection
3. Patient who admitted to any hospital in the Gulf and has Acute MI with confirm or suspicious of COVID-19 infection

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (1) Retrospective data for all patients since the COVID-19 appear in Qatar unit the prospective arm gets started after approval(2) Prospective data starting from the date of submission of this protocol and forward and all patients will be followed up for long-term outcome(3) Retrospective data for all cardiac patients hospitalizations in the COVID period of this year 2020 will be compared to previous years to report the trends of acute cardiovascular conditions in the COVID era to previous data, as a lot of countries documented decrease in the incidence.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The impact of COVID-19 on cardiovascular patient | 2 month from starting date
  The outcome of this registry will be:
  * entire information about the patients who admitted with COVID-19 accompany with a cardiovascular condition in Qatar.
  * Additionally, a comparison will be conducted between the cardiac patient who admitted over the period February to December to December 2020 and the same category of patients over the same period of 2019 in Qatar to figure out the reason behind the dropping of the number of the patient.
  * A multicenter data from the Gulf countries for Acute MI patients infected with COVID-19.
  * A comparison between our patients (either in Qatar only or the entire Gulf) populations and the outcome of other international registries such as the NACMI (US registry)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Jassim Alsuwaidi Senior Consultant, Principal Investigator — HMC
Locations (1):
- Hamad Medical Corporation, Doha, Unlisted (UL), Qatar